CLINICAL TRIAL: NCT00318058
Title: A Phase I/II, Open, Controlled Study in Order to Evaluate the Reactogenicity and the Immunogenicity of GlaxoSmithKline Biologicals Influenza Candidate Adjuvanted Vaccine in an Elderly Population Aged Over 65 Years Previously Vaccinated in 2004 With the Same Candidate Vaccine
Brief Title: Safety Study of an Adjuvanted Candidate Influenza Vaccine to Prevent Influenza Disease in the Elderly Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104540
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: influenza vaccine Fluarix, Adjuvanted Fluarix

SUMMARY:
As influenza vaccine efficacy is reported to be lower in elderly subjects compared to healthy adults, probably as a result of immunosenescence, there is a desire to devise ways to increase the current vaccines efficacy for this target population. Adjuvants are known to boost immune responses, thus representing one way to increase the efficacy of the current GlaxoSmithKline Fluarix™ influenza vaccine in elderly subjects. The purpose of this study is to evaluate the immunogenicity and the reactogenicity of a revaccination with the adjuvanted GlaxoSmithKline influenza vaccine administered intramuscularly about 1 year after administration of the first dose of vaccine. For immunogenicity and safety evaluations, subjects who have already received Fluarix™ during the preceeding year will receive a dose of commercial vaccine and will form the control group of this trial.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged over 65 years at the time of the revaccination; who previously received the adjuvanted candidate vaccine or Fluarix during a clinical study organized during the preceeding year

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* History of confirmed influenza infection since a year from the date of previous vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-10-03 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2005-11-04 (Actual)

PRIMARY OUTCOMES:
Percentage, intensity and relationship to vaccination of local (at the injection site) and general signs and symptoms during a 21 day follow-up period after vaccination
Occurrence of serious adverse events during the entire study.

SECONDARY OUTCOMES:
evaluation of the humoral immune response (haemagglutinin antibody titre) and cellular mediated immune response

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 104540 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/104540?search=study&#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104540 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register